CLINICAL TRIAL: NCT02877654
Title: Assessment of Intestinal Barrier in Irritable Bowel Syndrome Patients : Is There Any Correlation Between Plasmatic Zonulin and Expression of Intestinal Tight Junction Proteins ?
Brief Title: Is There Any Correlation Between Plasmatic Zonulin and Expression of Intestinal Tight Junction Proteins in IBS Patients?
Acronym: BISII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2015/174/HP
Record Dates: First submitted 2016-08-16; First posted 2016-08-24 (Estimated); Last update posted 2022-05-26 (Actual); Status verified 2021-09

CONDITIONS: Irritable Bowel Syndrome
Keywords: Plasmatic zonulin; Irritable Bowel Syndrome; Intestinal permeability
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Colonoscopy; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Irritable Bowel Syndrome (Experimental)
  Interventions: Procedure: colonoscopy with biopsies in the left colon to assess intestinal permeability

INTERVENTIONS:
Procedure: colonoscopy with biopsies in the left colon to assess intestinal permeability — Eleven colonic biopsies are taken in the left colon during colonoscopy. Intestinal permeability is assessed by western blot, qPCR and immunofluorescence for claudin; occludin and ZO-1.
  One blood sample is taken to assess plasmatic zonulin (ELISA kit).

SUMMARY:
Increased intestinal permeability is one of the main pathophysiological mechanisms involved in irritable bowel syndrome. The expression of some intestinal tight junction proteins is decreased mostly in IBS-diarrhoea patients. This decrease is correlated with increased intestinal permeability. Currently, no test used in clinical practice could assess intestinal permeability.

We hypothesis plasmatic zonulin could reflect intestinal permeability in IBS patients.

DETAILED DESCRIPTION:
The goal of our study is to look for a correlation between plasmatic zonulin and increased colonic permeability (assessed by the expression of intestinal tight junction proteins by western blot) in IBS patients and to look for a role of intestinal low-grade inflammation and microbiota.

Population :

IBS patients with diarrhoea or IBS with constipation or mixed with worsening of symptoms

Outcomes measures :

Plasmatic zonulin (ELISA kit) Occludin expression in colonic biopsies (western blot)

ELIGIBILITY:
Inclusion Criteria:

* IBS-Diarrhoea, IBS-constipation or alternating with recent worsening of symptoms, according to Rome III criteria
* Effective contraception since 1 month for women in childbearing age

Exclusion Criteria:

* Patients with organic and/or inflammatory digestive disease
* IBS with constipation or alternating without clinical warning sign
* Treatment such as anti-inflammatory, probiotic in the last three months
* Severe renal failure
* Hypersensitivity to Normacol
* Patient with blood dyscrasia disorder known or identified, anticoagulant or antiplatelet treatments
* Anal pathology (anal fissure, hemorrhoidal thrombosis)
* Pregnant or breastfeeding women
* Person with administrative or judicial decision or under legal protection measure
* Patient participating in another trial in the last two weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-05-20 (Actual)

PRIMARY OUTCOMES:
occludin level expression in left colonic biopsies | day 1
  occludin expression is measured using western blot (for proteins), q RT-PCT (for RNA) and IF (for localization).
  Plasmatic zonulin is measured in plasma using ELISA kit.
plasmatic zonulin expression | day 1
  Plasmatic zonulin expression is done using ELISA kit

SECONDARY OUTCOMES:
Claudin and ZO-1 level expression in left colonic biopsies | day 1
  Claudin and ZO-1 expression is measured using western blot (for proteins), q RT-PCT (for RNA) and IF (for localization)
Faecal calprotectin level | day 1
  Level is assessed on stool sample by ELISA kit in µg/g
Quality of life (GIQLI) | day 1
  Evaluation of quality of life using the validated score : french version of the Gastrointestinal Quality of Life Index (GIQLI).
Abdominal symptoms | day 1
  Abdominal symptoms of IBS are assessed with IBS symptom severity scale.
Anxiety and depression levels | day 1
  Anxiety and depression are assessed with the Hospital anxiety and depression scale.

CONTACTS AND LOCATIONS:
Overall Officials: Chloé Melchior, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No